CLINICAL TRIAL: NCT00003594
Title: A Randomized Phase III Trial of Three Different Regimens of CPT-11 Plus 5-Fluorouracil and Leucovorin Compared to 5-Fluorouracil and Leucovorin in Patients With Advanced Adenocarcinoma of the Colon and Rectum
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9741; CDR0000066665 (Registry Identifier: PDQ (Physician Data Query)); CAN-NCIC-CO13
Record Dates: First submitted 1999-11-01; First posted 2003-09-25 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- irinotecan + leucovorin + fluorouracil (Experimental): Patients receive irinotecan IV over 90 minutes followed by leucovorin calcium IV over 15 minutes and fluorouracil IV once a week for 4 weeks followed by 2 weeks of rest. Courses repeat every 6 weeks.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed before treatment, during treatment (arm specific), and after completion of treatment.
  Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.
  Interventions: Drug: irinotecan; Drug: fluorouracil; Drug: leucovorin calcium
- oxaliplatin + leucovorin + fluorouracil (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1 and leucovorin calcium IV over 2 hours plus fluorouracil IV over 22 hours on days 1 and 2. Courses repeat every 2 weeks.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed before treatment, during treatment (arm specific), and after completion of treatment.
  Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin
- oxaliplatin + irinotecan (Experimental): Patients receive oxaliplatin IV over 2 hours and irinotecan IV over 30 minutes on day 1. Courses repeat every 3 weeks.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed before treatment, during treatment (arm specific), and after completion of treatment.
  Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.
  Interventions: Drug: irinotecan; Drug: oxaliplatin

INTERVENTIONS:
Drug: irinotecan
  Arms: irinotecan + leucovorin + fluorouracil; oxaliplatin + irinotecan
Drug: fluorouracil
  Arms: irinotecan + leucovorin + fluorouracil; oxaliplatin + leucovorin + fluorouracil
Drug: leucovorin calcium
  Arms: irinotecan + leucovorin + fluorouracil; oxaliplatin + leucovorin + fluorouracil
Drug: oxaliplatin
  Arms: oxaliplatin + irinotecan; oxaliplatin + leucovorin + fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of combination chemotherapy is most effective in treating advanced colorectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of various combination chemotherapy regimens in treating patients who have advanced, recurrent, or metastatic colorectal cancer that cannot be treated with surgery or radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to progression in patients with locally advanced, locally recurrent, or metastatic colorectal adenocarcinoma treated with combinations of oxaliplatin, fluorouracil, leucovorin calcium, and irinotecan.
* Compare the quality of life, response rate, time to treatment failure, and overall survival in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to ECOG performance status (0-1 vs 2), prior adjuvant chemotherapy (yes vs no), prior immunotherapy (yes vs no), and age (under 65 vs 65 and over). Patients are randomized to one of three treatment arms.

Only arm II remains open to accrual.

* Arm I (Saltz regimen): Patients receive irinotecan IV over 90 minutes followed by leucovorin calcium IV over 15 minutes and fluorouracil IV once a week for 4 weeks followed by 2 weeks of rest. Courses repeat every 6 weeks. (Arm I closed to accrual as of March 15, 2002.)
* Arm II (FOLFOX4 regimen): Patients receive oxaliplatin IV over 2 hours on day 1 and leucovorin calcium IV over 2 hours plus fluorouracil IV over 22 hours on days 1 and 2. Courses repeat every 2 weeks.
* Arm III (oxaliplatin plus irinotecan): Patients receive oxaliplatin IV over 2 hours and irinotecan IV over 30 minutes on day 1. Courses repeat every 3 weeks. (Arm III closed to accrual as of March 15, 2002.) Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before treatment, during treatment (arm specific), and after completion of treatment.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 825 patients (275 per arm) have been accrued for this study thus far. Additional patients are being accrued on arm II. (Arms I and III closed to accrual as of March 15, 2002.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced, locally recurrent, or metastatic colorectal adenocarcinoma not curable by surgery or radiotherapy

  * Histological or cytological requirement waived in patients who developed radiological or clinical evidence of metastatic cancer after a prior surgical resection unless:

    * More than 5 years has elapsed since primary surgery OR
    * Primary cancer was stage I or II
* Site of primary lesion must be or have been confirmed endoscopically, radiologically, or surgically to be or have been in the large bowel
* Measurable or evaluable disease
* No CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL (transfusion allowed)

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No uncontrolled hypertension
* No unstable angina
* No symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* No serious uncontrolled arrhythmia
* No New York Heart Association class III or IV cardiac disease

Pulmonary:

* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* No pleural effusion or ascites that cause respiratory compromise (grade 2 or worse dyspnea)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active or uncontrolled infection
* No symptomatic sensory peripheral neuropathy
* No known allergy to platinum compounds
* No history of gastrointestinal bleeding unless it is determined to be acceptable by the enrolling physician
* No other prior or concurrent malignancy within the past 3 years except nonmelanoma skin cancer, carcinoma in situ of the uterine cervix, or other resected malignant tumor with less than a 10% probability of tumor relapse within 3 years of diagnosis
* No medical or psychiatric conditions that would preclude study
* No colonic or small bowel disorders with uncontrolled symptoms of more than 3 loose stools per day
* Colostomy or ileostomy allowed at investigator's discretion

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior adjuvant immunotherapy for resected stage II-IV disease allowed if adjuvant therapy concluded at least 1 year before documentation of recurrent disease
* No concurrent sargramostim (GM-CSF)

Chemotherapy:

* No prior chemotherapy for advanced colorectal cancer
* No prior standard adjuvant chemotherapy for rectal cancer
* Prior adjuvant fluorouracil for resected stage II-IV disease allowed if adjuvant therapy concluded at least 1 year before documentation of recurrent disease

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior major radiotherapy (e.g., chest or bone palliative radiotherapy)
* No prior radiotherapy to more than 15% of bone marrow
* No prior standard adjuvant radiotherapy for rectal cancer

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior major surgery (e.g., laparotomy) (2 weeks for minor surgery) and recovered
* Insertion of a vascular access device not considered major or minor surgery

Other:

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1691 (Actual)
Dates: Start 1998-10; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
time to progression | Up to 5 years

SECONDARY OUTCOMES:
overall survival | Up to 5 years
time to treatment failure | Up to 5 years
response rate | Up to 5 years
quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry C. Pitot, MD, Study Chair — Mayo Clinic
Locations (465):
- United States (429):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - Community Hospital of the Monterey Peninsula, Monterey, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University Medical Center, Stanford, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Columbia Medical Center of Aurora North Campus, Aurora, Colorado
  - Penrose Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian-St Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - HealthOne Rose Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Northern Colorado, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - Bristol Hospital, Bristol, Connecticut
  - University of Connecticut Health Center, Farmington, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - New Britain General Hospital, New Britain, Connecticut
  - Lawrence and Memorial Hospital, New London, Connecticut
  - William W. Backus Hospital, Norwich, Connecticut
  - Northwestern Connecticut Oncology-Hematology Associates, Torrington, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Florida - Gainesville, Gainesville, Florida
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - BroMenn Lifecare Center, Bloomington, Illinois
  - St. Joseph's Hospital Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Hematology Oncology Associates of Illinois - Lake Shore Dr, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Holy Family Medical Center, Des Plaines, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Northwest Oncology and Hematology, S.C., Elk Grove Village, Illinois
  - Eureka Hospital, Eureka, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex Hospital, Hopedale, Illinois
  - Silver Cross Hospital, Joliet, Illinois
  - Joliet Oncology/Hematology Associates, Ltd., Joliet, Illinois
  - Saint Joseph Medical Center, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Deerpath Medical Associates, Lake Forest, Illinois
  - North Shore Oncology Hematology Associates, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Hematology/Oncology Associates of Illinois, LLC, Melrose Park, Illinois
  - Mendota Community Hospital, Mendota, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Morris Hospital, Morris, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Hematology Oncology Associates of Illinois, LLC, Oak Park, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Affiliated Urology Specialists, Peoria, Illinois
  - Midwest Urological Group, Peoria, Illinois
  - Peoria Urological Associates, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Midwest Radiation Oncology Physicians, Peoria, Illinois
  - St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - St. James Hospital, Pontiac, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Trinity Medical Center, Rock Island, Illinois
  - Swedish-American Health System, Rockford, Illinois
  - Sarah D. Culbertson Memorial Hospital, Rushville, Illinois
  - Edward H. Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Midwest Cancer Research Group, Inc., Skokie, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Therapy Associates Hematology/Oncology, Evansville, Indiana
  - Oncology Institute of Greater Lafayette, Lafayette, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - William R. Bliss Cancer Center, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Medical Center, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Alegent Health Southwest Iowa Medical Center, Council Bluffs, Iowa
  - Des Moines General Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Mercy Cancer Center, Mason City, Iowa
  - Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Oncology & Hematology of Ottumwa, PC, Ottumwa, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Arkansas City, Arkansas City, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Radiation Oncology Center, Dodge City, Kansas
  - Halstead Cancer Center of Kansas, Halstead, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Liberal Cancer Center of Kansas, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Women's Health - Wichita, Wichita, Kansas
  - Wichita Clinic Cancer Medicine Associates, P.A., Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Faulkner Hospital, Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Lawrence Memorial Hospital of Medford/Hallmark Health Systems, Medford, Massachusetts
  - Morton Hospital & Medical Center, Taunton, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Genesee Regional Medical Center, Flint, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Office of E. Michael Lodish, Madison Heights, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - Balcueva Clinic, Saginaw, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria Clinic, Alexandria, Minnesota
  - Alexandria Radiation Oncology, Alexandria, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's/Duluth Clinic Health System, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, Fergus Falls, Minnesota
  - Mercy/Unity Hospitals, Fridley, Minnesota
  - Central Mesabi Medical Center, Hibbing, Minnesota
  - Duluth Clinic - Hibbing, Hibbing, Minnesota
  - Radiation Therapy Center, Hibbing, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - North Memorial Research Center, Minneapolis, Minnesota
  - Fairview University Medical Center - Riverside Campus, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Healtheast Cancer Care, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - Bryan LGH Medical Center, Lincoln, Nebraska
  - Prairie View Clinic, Lincoln, Nebraska
  - Bryan LGH Medical Center East, Lincoln, Nebraska
  - Office of Susan Hansen, M.D., Lincoln, Nebraska
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Wedgewood Medical Center, Lincoln, Nebraska
  - Southeast Nebraska Hematology, Lincoln, Nebraska
  - Southeast Nebreska Hematology-Oncology Consultants, PC, Lincoln, Nebraska
  - Williamsburg Radiation Oncology Center, Lincoln, Nebraska
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - Oncology Hematology West, P.C., Omaha, Nebraska
  - Alegent Health - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Cancer Center, Omaha, Nebraska
  - St. Joseph Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alegent Health-Midlands Community Hospital, Papillion, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Center for Cancer And Hematologic Disease, Cherry Hill, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Southern Oncology-Hematology Associates, P.A., Vineland, New Jersey
  - Comprehensive Cancer and Hematology Associates, Voorhees Township, New Jersey
  - Burlington County Hematology Oncology Association, P.A., Willingboro, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Health System, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Ireland Cancer Center, Canton, Ohio
  - Aultman Cancer Center, Canton, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - Woman Wise Blanchard Valley Regional Health Center, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Office of Sharon Cole, M.D., Kenton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - North West Ohio Oncology Center, Maumee, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - St. Charles Hospital, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Inc., Sandusky, Ohio
  - Flower Hospital - Pro Medica Health System, Sylvania, Ohio
  - Riverside Hospital, Toledo, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Hospital, Toledo, Ohio
  - MCO Cancer Institute, Toledo, Ohio
  - Haematology-Oncology Associates, Inc., Toledo, Ohio
  - Toledo Clinic, Inc., Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Muhlenberg Hospital Center, Bethlehem, Pennsylvania
  - Marion Community Hospital, Carbondale, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - DuBois Regional Medical Center, DuBois, Pennsylvania
  - UPMC Horizon, Greenville, Pennsylvania
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Wayne Memorial Hospital, Honesdale, Pennsylvania
  - UPCI @ UPMC Lee Hospital, Johnstown, Pennsylvania
  - Conemaugh Memorial Hospital, Johnstown, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Regional Center, Langhorne, Pennsylvania
  - Latrobe Area Hospital, Latrobe, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, Lemoyne, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC/Passavant Hospital, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Moses Taylor Hospital, Scranton, Pennsylvania
  - Scranton Hematology-Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sioux Valley Clinic, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital, Sioux Falls, South Dakota
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Memorial Medical Center, Ashland, Wisconsin
  - Luther Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic, Eau Claire, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - Dean Medical Center, Madison, Wisconsin
  - Meriter Hospital, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Aurora Sinai Samaritan Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center Wausau Hospital, Wausau, Wisconsin
- Canada (31):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Nanaimo Cancer Clinic, Nanaimo, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Algoma District Medical Group, Sault Ste. Marie, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - CHUM Hopital Saint-Luc, Montreal, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Lions Gate Hospital, North Vancouver
- Puerto Rico (3):
  - Centro Mamografia Hospital Oncologico, Hato Rey
  - Veterans Affairs Medical Center - San Juan, San Juan
  - San Juan City Hospital, San Juan
- South Africa (2):
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Pretoria Academic Hospitals, Pretoria

REFERENCES:
- [Background] Franko J, Shi Q, Goldman CD, Pockaj BA, Nelson GD, Goldberg RM, Pitot HC, Grothey A, Alberts SR, Sargent DJ. Treatment of colorectal peritoneal carcinomatosis with systemic chemotherapy: a pooled analysis of north central cancer treatment group phase III trials N9741 and N9841. J Clin Oncol. 2012 Jan 20;30(3):263-7. doi: 10.1200/JCO.2011.37.1039. Epub 2011 Dec 12. PMID 22162570
- [Background] An MW, Mandrekar SJ, Branda ME, Hillman SL, Adjei AA, Pitot HC, Goldberg RM, Sargent DJ. Comparison of continuous versus categorical tumor measurement-based metrics to predict overall survival in cancer treatment trials. Clin Cancer Res. 2011 Oct 15;17(20):6592-9. doi: 10.1158/1078-0432.CCR-11-0822. Epub 2011 Aug 31. PMID 21880789
- [Background] Campbell ME, Mandrekar SJ, Hillman SL, et al.: What is the added value of actual tumor measurements (TM) in predicting overall survival (OS)? The North Central Cancer Treatment Group (NCCTG) findings. [Abstract] J Clin Oncol 26 (Suppl 15): A-6520, 2008.
- [Background] Grothey A, Hedrick EE, Mass RD, Sarkar S, Suzuki S, Ramanathan RK, Hurwitz HI, Goldberg RM, Sargent DJ. Response-independent survival benefit in metastatic colorectal cancer: a comparative analysis of N9741 and AVF2107. J Clin Oncol. 2008 Jan 10;26(2):183-9. doi: 10.1200/JCO.2007.13.8099. PMID 18182660
- [Background] Grothey A, Hedrick EE, Mass RD, et al.: Response rate using conventional criteria is a poor surrogate for clinical benefit on progression-free (PFS) and overall survival (OS) in metastatic colorectal cancer (mCRC): a comparative analysis of N9741 and AVF2107. [Abstract] J Clin Oncol 24 (Suppl 18): A-3516, 2006.
- [Background] Goldberg R. Oxaliplatin in colorectal cancer: current studies. Oncology (Williston Park). 2000 Dec;14(12 Suppl 11):42-7. PMID 11204663
- [Result] Heun JM, Grothey A, Branda ME, Goldberg RM, Sargent DJ. Tumor status at 12 weeks predicts survival in advanced colorectal cancer: findings from NCCTG N9741. Oncologist. 2011;16(6):859-67. doi: 10.1634/theoncologist.2011-0064. Epub 2011 May 31. PMID 21632455
- [Result] Ng K, Sargent DJ, Goldberg RM, Meyerhardt JA, Green EM, Pitot HC, Hollis BW, Pollak MN, Fuchs CS. Vitamin D status in patients with stage IV colorectal cancer: findings from Intergroup trial N9741. J Clin Oncol. 2011 Apr 20;29(12):1599-606. doi: 10.1200/JCO.2010.31.7255. Epub 2011 Mar 21. PMID 21422438
- [Result] Goldberg RM, Sargent DJ, McLeod H. Leveraging learning from a phase III colorectal cancer clinical trial: outcomes, methodology, meta-analysis and pharmacogenetics. Trans Am Clin Climatol Assoc. 2010;121:21-32; discussion 32-3. PMID 20697547
- [Result] McLeod HL, Sargent DJ, Marsh S, Green EM, King CR, Fuchs CS, Ramanathan RK, Williamson SK, Findlay BP, Thibodeau SN, Grothey A, Morton RF, Goldberg RM. Pharmacogenetic predictors of adverse events and response to chemotherapy in metastatic colorectal cancer: results from North American Gastrointestinal Intergroup Trial N9741. J Clin Oncol. 2010 Jul 10;28(20):3227-33. doi: 10.1200/JCO.2009.21.7943. Epub 2010 Jun 7. PMID 20530282
- [Result] Goldberg RM, Sargent DJ, Morton RF, Green E, Sanoff HK, McLeod H, Buckner J. NCCTG Study N9741: leveraging learning from an NCI Cooperative Group phase III trial. Oncologist. 2009 Oct;14(10):970-8. doi: 10.1634/theoncologist.2009-0175. Epub 2009 Oct 14. PMID 19828593
- [Result] Sanoff HK, Sargent DJ, Green EM, McLeod HL, Goldberg RM. Racial differences in advanced colorectal cancer outcomes and pharmacogenetics: a subgroup analysis of a large randomized clinical trial. J Clin Oncol. 2009 Sep 1;27(25):4109-15. doi: 10.1200/JCO.2009.21.9527. Epub 2009 Jul 27. PMID 19636001
- [Result] Fuchs CS, Goldberg RM, Sargent DJ, Meyerhardt JA, Wolpin BM, Green EM, Pitot HC, Pollak M. Plasma insulin-like growth factors, insulin-like binding protein-3, and outcome in metastatic colorectal cancer: results from intergroup trial N9741. Clin Cancer Res. 2008 Dec 15;14(24):8263-9. doi: 10.1158/1078-0432.CCR-08-0480. Epub 2008 Dec 10. PMID 19073970
- [Result] Sanoff HK, Sargent DJ, Campbell ME, Morton RF, Fuchs CS, Ramanathan RK, Williamson SK, Findlay BP, Pitot HC, Goldberg RM. Five-year data and prognostic factor analysis of oxaliplatin and irinotecan combinations for advanced colorectal cancer: N9741. J Clin Oncol. 2008 Dec 10;26(35):5721-7. doi: 10.1200/JCO.2008.17.7147. Epub 2008 Nov 10. PMID 19001325
- [Result] Sargent DJ, Campbell M, Grothey A, et al.: Overall and 12 week tumor response versus actual tumor measurements as predictors of overall survival (OS) in advanced colorectal cancer (ACRC): findings from NCCTG N9741. [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-446, 2008.
- [Result] Dy GK, Krook JE, Green EM, Sargent DJ, Delaunoit T, Morton RF, Fuchs CS, Ramanathan RK, Williamson SK, Findlay BP, Pockaj BA, Sticca RP, Alberts SR, Pitot HC 4th, Goldberg RM; Intergroup N9741. Impact of complete response to chemotherapy on overall survival in advanced colorectal cancer: results from Intergroup N9741. J Clin Oncol. 2007 Aug 10;25(23):3469-74. doi: 10.1200/JCO.2007.10.7128. PMID 17687151
- [Result] Grothey A, Sargent DJ, Campbell ME, et al.: Waterfall plots provide detailed information on magnitude of response to conventional chemotherapy in colorectal cancer: lessons learned from N9741. [Abstract] American Society of Clinical Oncology 2007 Gastrointestinal Cancers Symposium, 19 -21 January 2007, Orlando, Florida A-337, 2007.
- [Result] Goldberg RM, McLeod HL, Sargent DJ, et al.: Genetic polymorphisms, toxicity, and response rate in African Americans (AA) with metastatic colorectal cancer (MCRC) compared to Caucasians (C) when treated with IFL, FOLFOX or IROX in Intergroup N9741. [Abstract] J Clin Oncol 24 (Suppl 18): A-3503, 2006.
- [Result] Goldberg RM, Sargent DJ, Morton RF, Fuchs CS, Ramanathan RK, Williamson SK, Findlay BP, Pitot HC, Alberts S. Randomized controlled trial of reduced-dose bolus fluorouracil plus leucovorin and irinotecan or infused fluorouracil plus leucovorin and oxaliplatin in patients with previously untreated metastatic colorectal cancer: a North American Intergroup Trial. J Clin Oncol. 2006 Jul 20;24(21):3347-53. doi: 10.1200/JCO.2006.06.1317. PMID 16849748
- [Result] McLeod HL, Parodi L, Sargent DJ, et al.: UGT1A1*28, toxicity and outcome in advanced colorectal cancer: results from trial N9741. [Abstract] J Clin Oncol 24 (Suppl 18): A-3520, 2006.
- [Result] Delaunoit T, Alberts SR, Sargent DJ, Green E, Goldberg RM, Krook J, Fuchs C, Ramanathan RK, Williamson SK, Morton RF, Findlay BP. Chemotherapy permits resection of metastatic colorectal cancer: experience from Intergroup N9741. Ann Oncol. 2005 Mar;16(3):425-9. doi: 10.1093/annonc/mdi092. Epub 2005 Jan 27. PMID 15677624
- [Result] Dy GK, Krook J, Green E, et al.: Impact of complete response to chemotherapy on overall survival (OS) in advanced colorectal cancer (CRC): results from Intergroup N9741. [Abstract] American Society of Clinical Oncology 2005 Gastrointestinal Cancers Symposium, 27-29 January 2005, Miami, Florida. A-185, 2005.
- [Result] Delaunoit T, Goldberg RM, Sargent DJ, Morton RF, Fuchs CS, Findlay BP, Thomas SP, Salim M, Schaefer PL, Stella PJ, Green E, Mailliard JA. Mortality associated with daily bolus 5-fluorouracil/leucovorin administered in combination with either irinotecan or oxaliplatin: results from Intergroup Trial N9741. Cancer. 2004 Nov 15;101(10):2170-6. doi: 10.1002/cncr.20594. PMID 15470715
- [Result] Goldberg RM, Sargent DJ, Morton RF, Fuchs CS, Ramanathan RK, Williamson SK, Findlay BP, Pitot HC, Alberts SR. A randomized controlled trial of fluorouracil plus leucovorin, irinotecan, and oxaliplatin combinations in patients with previously untreated metastatic colorectal cancer. J Clin Oncol. 2004 Jan 1;22(1):23-30. doi: 10.1200/JCO.2004.09.046. Epub 2003 Dec 9. PMID 14665611
- [Result] Goldberg RM, Morton RF, Sargent DJ, et al.: N9741: oxaliplatin (Oxal) or CPT-11 + 5-fluorouracil (5FU)/leucovorin (LV) or oxal + CPT-11 in advanced colorectal cancer (CRC). Updated efficacy and quality of life (QOL) data from an intergroup study. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1009, 252, 2003.
- [Result] Goldberg RM, Morton RF, Sargent D, et al.: N9741: oxaliplatin (oxal) or CPT-11 + 5-fluorouracil (5FU)/leucovorin (LV) or oxal + CPT-11 in advanced colorectal cancer (CRC). Initial toxicity and response data from a GI Intergroup study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-511, 2002.
- [Result] Morton RF, Goldberg RM, Sargent DJ, et al.: Oxaliplatin (OXAL) or CPT-11 Combined with 5FU/Leucovorin (LV) in Advanced Colorectal Cancer (CRC): an NCCTG/CALGB Study. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-495, 2001.
- [Derived] Yuan C, Renfro L, Ambadwar PB, Ou FS, McLeod HL, Innocenti F, Meyerhardt JA, Wolpin BM, Goldberg RM, Grothey A, Fuchs CS, Ng K. Influence of genetic variation in the vitamin D pathway on plasma 25-hydroxyvitamin D3 levels and survival among patients with metastatic colorectal cancer. Cancer Causes Control. 2019 Jul;30(7):757-765. doi: 10.1007/s10552-019-01183-1. Epub 2019 May 18. PMID 31104167
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/